CLINICAL TRIAL: NCT04408950
Title: Sample Collection for Systems Evaluation of Patients With Unknown or Incompletely Characterized Immune Defects
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200084; 20-I-0084
Record Dates: First submitted 2020-05-29; First posted 2020-06-01 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11-17

CONDITIONS: Immunodeficiency
Keywords: Immunological Disorders; Monogenic; Systems Immunology; Phenotype; Hypothesis Generating; Natural History
MeSH Terms: conditions — Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with uncharacterized immune defects: Patients with uncharacterized immune defects
- Unaffected biological relatives: Unaffected biological relatives

SUMMARY:
Background:

The immune system defends the body against disease. It has many different parts spread out in

the body, including in the blood and skin. To learn more about it, researchers want to study samples from people with healthy immune systems and people with conditions that affect how the immune system works.

Objective:

To learn about how the different parts of the immune system come together to make a whole.

Eligibility:

People age 2 and older who have a condition that affects the immune system or have a family member with such a condition.

Design:

Participants will be screened with medical and medicine review. Other lab tests may also be reviewed. Some participants will take a pregnancy test.

Participants will give blood samples. They may also give saliva, stool, and urine samples.

A sterile cotton swab may be rubbed over their skin or inside the cheek or nose to collect cells.

If participants have samples collected as part of their regular medical care, their doctor may be asked to send parts of the samples that otherwise would be thrown away. These samples may be from biopsies, endoscopies, or other procedures.

Some participants may have optional skin punch biopsies. For this, their skin is numbed. Then a tool removes 1 or 2 small pieces of skin from the forearm or thigh.

Participants medical records will be checked to see if they have any changes in their health over time. If they have a study visit, they may talk about their medical history and have a physical exam.

Participation lasts 5 years....

DETAILED DESCRIPTION:
Immunological disorders predispose affected individuals to a myriad of complications, including infection, immune dysregulation with autoimmune disease and aberrant inflammatory responses, and malignancy. Advances in genetic testing have propelled the discovery of the genetic underpinnings of numerous immunodeficiencies. However, a more complete picture of the immune system is needed to better characterize patients that present with the signs and symptoms of immunodeficiency or immune dysregulation in whom there is no identifiable genetic diagnosis. Many of our diagnostic tools, such as characterization of cell subset frequencies, look at only one parameter in the immune system, which is typically insufficient to capture the system s complexity. Systems immunology is a field of research aimed to identify and understand how the different components of the immune system work together in a coordinated manner to achieve its functions, such as protecting against pathogens and mounting effective responses after vaccination. The goal of this study is to collect patient samples to more deeply phenotype these individuals at the molecular and cellular levels using novel technologies in order to generate hypotheses regarding disease etiologies and mechanisms in subjects with an immune disorder without complete characterization or clear genetic etiology. We also aim to validate a specific observation seen in a previous study of patients with known monogenic immunological disorders. In the long-term, hypotheses generated in this study that address clinically significant, actionable questions will be pursued as separate investigations.

This hypothesis-generating sample collection study will recruit patients with unknown or incompletely characterized immune defects and their unaffected relatives. Under this protocol, samples will be collected at the NIH Clinical Center or mailed in for analysis using systems biology approaches to generate hypotheses regarding the potential etiologies and mechanisms of these immune defects. Initially, all subjects will give a blood sample and may give additional samples including saliva, stool, and skin punch biopsies. Subjects will be enrolled for 5 years and may be asked to give additional samples based on scientific need or changes in clinical status. Findings relevant to subjects health and medical care will be returned to them and referring healthcare providers.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Aged greater than or equal to 2 years.
  2. Meets 1 of the following criteria:

     a. Patient with a suspected or known/molecularly defined but incompletely characterized immune disorder (as determined by a referring NIH study staff member) AND meeting at least one of the following:

     i. within 1 year of screening, abnormal immune function demonstrated by at least one laboratory test result outside the normal range

     ii. history of severe or atypical infection, immune dysregulation (defined as autoimmunity, lymphoproliferation, or HLH), or autoinflammatory symptoms (defined as episodic fever often associated with dermatitis, gastrointestinal symptoms, and arthropathy).

     b. Biological unaffected relative of an individual meeting criterion 2a but who does not meet criterion 2a himself/herself. Unaffected relatives may be mother, father, siblings, children, grandparents, aunts, uncles, or first cousins to the individual.
  3. Willing to allow storage of samples and data for future research.
  4. For patients, currently or previously enrolled on an NIH protocol that performs WES or WGS and that allows sharing of sequence data.
  5. For unaffected relatives, able to provide informed consent.

EXCLUSION CRITERIA:

Individuals meeting any of the following criteria will be excluded from study participation:

1. History of secondary causes of immunodeficiency or dysregulation (e.g., HIV infection, immunodeficiency from chronic use of immunosuppressive or chemotherapeutic agents), at the discretion of the investigator.
2. Pregnancy.
3. Any condition that, in the opinion of the investigator, contraindicates participation in this study.

Ages: 2 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants will be selected or referred to the protocol from other NIH groups whose patients have an uncharacterized immune defect. Unaffected biological relatives of these participants may also be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
CBC with differential, lymphocyte phenotyping, and whole blood RNA expression data analyzed in individuals with unknown or incompletely characterized immune defects. | Baseline
  CBC with differential, lymphocyte phenotyping, and whole blood RNA expression data analyzed in individuals with unknown or incompletely characterized immune defects.

SECONDARY OUTCOMES:
CBC with differential and lymphocyte phenotyping in individuals with unknown or incompletely characterized immunological defects compared with age- and gender-matched healthy control | Baseline
  CBC with differential and lymphocyte phenotyping in individuals with unknown or incompletely characterized immunological defects compared with age- and gender-matched healthy control

CONTACTS AND LOCATIONS:
Overall Officials: Irini Sereti, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-I-0084.html